CLINICAL TRIAL: NCT02416661
Title: Lyso-Gb1 as a Long-term Prognostic Biomarker in Gaucher Disease: An International, Multicenter, Epidemiological Protocol
Brief Title: Lyso-Gb1 as a Long-term Prognostic Biomarker in Gaucher Disease
Acronym: LYSO-PROOF
Status: Completed | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: LP 06-2018
Record Dates: First submitted 2015-03-13; First posted 2015-04-15 (Estimated); Last update posted 2021-05-28 (Actual); Status verified 2020-04

CONDITIONS: Lysosomal Storage Diseases; Gaucher Disease; Sphingolipidoses
Keywords: Gaucher Disease type 1; Lymphatic Diseases; Lipid Metabolism, Inborn Errors; Lipid Metabolism Disorders; Lipidoses
MeSH Terms: conditions — Lysosomal Storage Diseases; Gaucher Disease; Sphingolipidoses; Lymphatic Diseases; Lipid Metabolism, Inborn Errors; Lipid Metabolism Disorders; Lipidoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample applied on the Dry Blood Spot (DBS) Filtercard (Centocard®)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Participants diagnosed with Gaucher disease: Participants with genetically confirmed diagnosis of Gaucher disease type 1 older than 6 months old

SUMMARY:
International, multicenter, epidemiological study to demonstrate the correlation and predictive value of lyso-Gb1 concentration with the clinical severity of naïve, initially non-ERT/SRT Gaucher disease type 1 and during the study ERT/SRT-newly started Gaucher type 1 patients and to correlate lyso-Gb1 concentration with the clinical improvement of ERT or SRT treated Gaucher type 1 and the clinical course of non-treated patients based on GD-DS3

DETAILED DESCRIPTION:
Gaucher disease is an autosomal recessive inherited lysosomal storage disorder. The disease is caused by the hereditary deficiency of the glucocerebrosidase, a lysosomal enzyme that breaks down glucocerebroside into glucose and ceramide.

To date a definitive diagnosis of Gaucher's disease can only be made applying biochemical testing measuring the reduced enzymatic activity of the beta-glucosidase together with genetic confirmation. Since numerous different mutations may be the cause of a particular lysosomal storage disease the sequencing of the entire beta-glucosidase gene is applied in Gaucher's disease in order to confirm the genetic diagnosis.

The use of primary storage molecules as biomarker was assessed for glucosylceramide (Gb1) in plasma of Gaucher's disease patients and compared to the level of Gb1 in healthy individuals.

In order to establish a sensitive and specific biomarker for GD, we compared mass spectra of the plasma of healthy controls and GD patients using HPLC and tandem mass spectrometry. Mass spectra that differed most between patients and controls were analysed in more detail. The resulting biomarker, which was patented in June 2011 (PCT/EP2012/002409), was lyso - Gb1. We identified this compound as a reliable, sensitive and specific biomarker for GD in a cohort of GD patients. Furthermore, in a pilot study we evaluated whether lyso-Gb1 is related to the specific genotypes and is reliable for long-term monitoring of the efficiency of therapy.

The aim this study is therefore to investigate lyso-Gb1 as a long-term prognostic marker in naïve, non-ERT/SRT GD type 1 patients by monitoring over the course of 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 6 months or older
* Patients with genetically confirmed diagnosis of Gaucher disease type 1
* No prior treatment with enzyme replacement therapy or substrate reduction therapy ro no traetment for more than 24 months
* Signed informed consent by parents/legal guardian and patient

Exclusion Criteria:

* Male or female patients being younger than 6 months
* Patients without genetically confirmed diagnosis of Gaucher disease type 1
* Gaucher disease 2 or 3
* Patient is currently undergoing enzyme replacement therapy or substrate reduction therapy
* Missing signed informed consent

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female patients aged 6 months or older with genetically confirmed diagnosis of Gaucher disease type 1 without treatment prior to enrollment or no treatment for more than 24 months ago
Sampling Method: Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Demonstrating the correlation and predictive value of lyso-Gb1 concentration with the clinical severity of naïve, initially non-ERT/SRT Gaucher disease type 1 and during the study ERT/SRT-newly started Gaucher type 1 patients | 48 month
  lyso-Gb1 will be analzyed via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS) and compared to merged control. The LC/MRM-MS is performed on an ABSciex 6500 triple quadrupole mass spectrometer, coupled with a Waters Acquity UPLC.

SECONDARY OUTCOMES:
Correlating lyso-Gb1 concentration with the clinical improvement of ERT or SRT treated Gaucher type 1 and the clinical course of non-treated patients based on GD-DS3. | 48 month
  lyso-Gb1 will be analysed over a period of 36 months via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS) to demonstrate the course of the biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, M.D., Study Chair — CENTOGENE GmbH Rostock
Locations (8):
- University Hospital Center Mother Teresa, Tirana, Albania
- Aristotle University of Thessaloniki, Ippokration General Hospital, Thessaloniki, Greece
- Centre for Human Genetics, Bangalore, India
- Shaare Zedek Medical Center, Jerusalem, Israel
- Morocco (2):
  - Children hospital, Rabat
  - Hopital d'Enfant, Rabat
- The Children's Hospital and the Institute of Child Health, Lahore, Punjab Province, Pakistan
- Hospital Universitari de Bellvitge (planta 7.1), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Elstein D, Mellgard B, Dinh Q, Lan L, Qiu Y, Cozma C, Eichler S, Bottcher T, Zimran A. Reductions in glucosylsphingosine (lyso-Gb1) in treatment-naive and previously treated patients receiving velaglucerase alfa for type 1 Gaucher disease: Data from phase 3 clinical trials. Mol Genet Metab. 2017 Sep;122(1-2):113-120. doi: 10.1016/j.ymgme.2017.08.005. Epub 2017 Aug 24. PMID 28851512